CLINICAL TRIAL: NCT07182370
Title: Polyphenol Metabolism and Personalized Nutrition in Menopause: Metabotypes, Microbiome-virome, and Relationship With Quality of Life and Cardiovascular Risk.
Brief Title: Polyphenol Metabolism and Personalized Nutrition in Menopause (PolyPause).
Acronym: PolyPause
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Hospital Universitario Virgen de la Arrixaca (Other); IMDEA Food (Other)
Responsible Party: Principal Investigator, Juan Carlos Espín de Gea, Full Research Professor, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PID2022-136419OB-I00
Record Dates: First submitted 2025-09-02; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Menopause Related Conditions; Cardiovascular Risk
Keywords: Menopause; Microbiome; Phageome; Cardiovascular risk; Gut dysbiosis; Quality of life; LDLox; TMAO; Bile acids; Blood lipids; resveratrol; pomegranate; urolithin; isoflavones; equol; Metabotype; Personalized nutrition; Lunularin; Ellagic acid; Endotoxemia; Short-chain farry acids
MeSH Terms: conditions — Endotoxemia | interventions — Ellagic Acid; Isoflavones

STUDY DESIGN:
Intervention Model Description: Crossover Assignment. Randomized, double-blind, placebo-controlled and crossover trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Polyphenol-rich capsules (PPs-A) (Experimental): Consumption of polyphenol-rich plant extrats (PPs).
  Interventions: Dietary Supplement: Capsules containing plant extracts, including resveratrol, ellagic acid and isoflavones
- (Placebo-A) (Placebo Comparator): Consumption of microcrystalline cellulose (placebo).
  Interventions: Dietary Supplement: Consumption of placebo
- Polyphenol-rich capsules (PPs-B) (Experimental): Consumption of polyphenol-rich plant extracts (PPs).
  Interventions: Dietary Supplement: Capsules containing plant extracts, including resveratrol, ellagic acid and isoflavones
- (Placebo-B) (Placebo Comparator): Consumption of microcrystalline cellulose (placebo).
  Interventions: Dietary Supplement: Consumption of placebo

INTERVENTIONS:
Dietary Supplement: Capsules containing plant extracts, including resveratrol, ellagic acid and isoflavones — Eight-week intake of three capsules per day, containing a total of 2.1 g of plant extracts (PPs), including 150 mg of resveratrol (found in grapes and red wine), 100 mg of ellagic acid (present in strawberries, walnuts, pomegranate, etc.), and 50 mg of the isoflavone daidzein, among others (found in soy, red clover, etc.).
  Arms: Polyphenol-rich capsules (PPs-A); Polyphenol-rich capsules (PPs-B)
Dietary Supplement: Consumption of placebo — Daily intake of three capsules (2.1 g/day) of microcrystalline cellulose for eight weeks
  Arms: (Placebo-A); (Placebo-B)

SUMMARY:
The study aims to evaluate the role of the gut microbiome and phageome in explaining interindividual variability in the metabolic response to polyphenol-rich nutraceuticals among menopausal women. Insights from this research will support the development of personalized nutrition strategies to improve quality of life and reduce cardiovascular disease (CVD) risk during menopause.

DETAILED DESCRIPTION:
This trial aims to investigate the role of the gut microbiome and phageome in mediating interindividual variability in the metabolic response to polyphenol-rich plant extracts among postmenopausal women. Polyphenols are widely recognized for their potential benefits in cardiovascular health, cognitive function, and overall metabolic regulation. However, the magnitude and direction of their effects vary significantly between individuals. Mounting evidence suggests that the gut microbiota plays a critical role in the biotransformation of polyphenols into bioactive metabolites, giving rise to the so-called gut microbiota metabotypes (i.e., metabolic fingerprints of the gut microbiota that produce specific metabolites depending on the individual), thereby modulating the physiological effects of ingested polyphenols.

A cohort of postmenopausal women will be studied at four timepoints in a randomized, double-blind, placebo-controlled, crossover trial. Participants will undergo a controlled dietary intervention with standardized polyphenol-rich plant extracts (pomegranate, soy, and resveratrol). The primary outcome will be a ≥15% change in serum oxidized LDL (oxLDL). At each timepoint, gut microbiome and phageome profiles will be characterized using shotgun metagenomic sequencing. TMAO, bile acids, and short-chain fatty acids will be determined by UPLC-QTOF-MS and GC-MS. Additional biomarkers of cardiovascular and metabolic health will be determined, including serum total cholesterol, LDLc, HDLc, and LPS-binding protein (LBP); fecal microbial enzymatic activities (β-glucuronidase and sulfatase); and serum neurotransmitters (GABA, dopamine, serotonin, melatonin, epinephrine, norepinephrine).

The distribution of polyphenol metabotypes in this cohort will be assessed through circulating and urinary phenolic-derived metabolites. This will allow exploration of differential individual responses to polyphenol intake and their derived health effects. Untargeted urinary metabolomics will further explore potential changes in metabolites relevant to cardiovascular prevention. Quality of life will be evaluated using the validated Cervantes Scales, which include domains related to menopause-associated symptoms, cognitive issues, and overall health.

The study is designed to integrate multi-omic data, combining microbial and phageomic composition with metabolomic and biochemical readouts, to identify patterns and predictors of individual responses to polyphenol intake. Statistical and bioinformatic analyses will focus on associations between microbiome/phageome signatures and metabolic outcomes, aiming to elucidate the mechanisms by which gut microbes and their viruses influence polyphenol biotransformation and subsequent systemic effects. This study therefore seeks to advance precision nutrition strategies for postmenopausal women. Insights gained may inform personalized dietary recommendations aimed at enhancing cardiovascular health, metabolic regulation, and overall quality of life during menopause. Moreover, the inclusion of the phageome represents a highly innovative and largely unexplored aspect of the study, offering new avenues for microbiota-targeted interventions.

Overall, this research will contribute to understanding the complex interactions between diet, the gut ecosystem, and human metabolism, ultimately supporting the development of evidence-based, individualized nutritional strategies to reduce cardiovascular disease risk and improve health outcomes in the postmenopausal population.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45 to 57 years.
* Diagnosed menopause (defined as 12 consecutive months without menstruation).
* Presenting at least one climacteric symptom (hot flashes and/or sweating episodes and/or low mood and/or irritability and/or decreased libido and/or insomnia and/or joint/muscle pain).
* Body Mass Index (BMI) ≥ 18 kg/m².
* Adequate cultural level and ability to understand the clinical study.
* Willing to voluntarily participate in the study and provide written informed consent.

Exclusion Criteria:

* Presence of severe, chronic-degenerative, or psychiatric conditions, or any contraindication to the use of nutritional supplements.
* History of major gastrointestinal surgery.
* Swallowing difficulties (e.g., inability to ingest capsules).
* BMI < 18 kg/m² or > 30 kg/m².
* Currently following a weight-loss regimen.
* Known or suspected allergy or intolerance to red clover extract, resveratrol (grape, wine), soy, or pomegranate.
* Use of chronic preventive medication for cholesterol, glucose, blood pressure, etc. (e.g., statins, metformin, beta-blockers).
* Use of antibiotics within one month prior to study initiation.
* Undergoing hormone replacement therapy.
* Alcohol consumption exceeding 1 beer or 1 glass of wine per day.
* Regular use of dietary supplements (e.g., probiotics, isoflavones, resveratrol, others).
* Following a vegetarian diet.
* Current smoker or having smoked at any time during the past year.
* Individuals unwilling to comply with study guidelines.

Ages: 45 Years to 57 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only individuals assigned female at birth who self-identify as women are eligible to participate, provided they meet the biological criteria for postmenopause as defined in the study protocol. While gender identity is fully respected, eligibility is determined by biological sex due to the physiological nature of the condition under investigation.
Enrollment: 90 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Oxidized LDL particles (LDLox) | Change from baseline at 8 weeks compared to placebo
  15% change in serum oxidized LDL concentration (U/L) by ELISA

SECONDARY OUTCOMES:
Gut microbiome | Change from baseline at 8 weeks compared to placebo
  Change in gut microbiome composition, including taxonomic relative abundance and α- and β-diversity indices, by shotgun metagenomic sequencing
Gut phageome | Change from baseline at 8 weeks compared to placebo
  Change in gut phageome composition, including taxonomic relative abundance and α- and β-diversity indices, by shotgun metagenomic sequencing
Blood lipids | Change from baseline at 8 weeks compared to placebo
  Change in serum total cholesterol, LDLc and HDLc concentration (mg/dL) by autoanalyzer
Trimethylamine N-oxide (TMAO) | Change from baseline at 8 weeks compared to placebo
  Change in serum (µM) and urine (µM/mg creatinine) TMAO concentration by UPLC-QTOF-MS
Lipopolysaccharide binding protein (LBP) | Change from baseline at 8 weeks compared to placebo
  Change in serum LBP concentration (µg/ml) by ELISA
Quality of life (Cervantes Scale) | Change from baseline at 8 weeks compared to placebo
  Changes in the domains of the Cervantes Scale (validated questionnaires): Health, psychological, sexuality, and couple relationship.
Short-chain fatty acids (SCFAs) | Change from baseline at 8 weeks compared to placebo
  Change in fecal SCFA concentration (µM/g) by GC-MS
Bile acids (BAs) | Change from baseline at 8 weeks compared to placebo
  Change in fecal BA concentration (µM/g) by UPLC-QTOF-MS
Change in serum neurotransmitters | Change from baseline at 8 weeks compared to placebo
  Change in serum gamma-aminobutyric acid (GABA, µM), serotonin, melatonin, dopamine, epinephrine, and norepinephrine (nM) by UPLC-QTOF-MS
Untargeted metabolomics | Change from baseline at 8 weeks compared to placebo
  Change in urinary metabolite concentrations (µg/mg creatinine) by UPLC-QTOF-MS
Gut microbiota metabotypes | Identification at baseline and after 8 weeks consuming the polyphenol-rich plant extracts
  Distribution of urolithin, equol, and resveratrol metabotypes in postmenopausal women by UPLC-QTOF-MS metabolite profiling
Estrobolome activity | Change from baseline at 8 weeks compared to placebo
  Change in fecal microbial glucuronidase and sulfatase activities (U/mg protein) by spectrophotometry

CONTACTS AND LOCATIONS:
Overall Officials: Juan C. Espín, PhD, Principal Investigator — Spanish National Research Council
Locations (1):
- Centro de Edafología y Biología Aplicada del Segura (CEBAS-CSIC), Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results (including raw metabolomics datasets from UPLC-QTOF-MS and GC-MS, and raw microbiome/phageome sequencing data) will be available upon reasonable request. Data will be shared after publication of the primary outcomes and will require a data use agreement to ensure appropriate use.
Supporting Information: Study Protocol
Time Frame: Time Frame: Beginning 12 months after publication of the results; available for 5 years.
Access Criteria: Access Criteria: Qualified researchers may request access by contacting the Principal Investigator. Data will be shared in a controlled manner to ensure confidentiality of participants.